CLINICAL TRIAL: NCT02898896
Title: Asymptomatic Obstructive Coronary Artery Disease (CAD) in Suppressed HIV-infected Patients ≥ 45 Years and 2 or More CV Risk Factors. Associations With Persistent Immune Activation and Microbial Translocation
Brief Title: Coronary Artery Disease (CAD) in Suppressed HIV-infected
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Departure of the coordinating investigator
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Hospital Universitario La Paz (Other); Hospital Reina Sofia, Murcia (Unknown); Hospital Vall D' Hebron Barcelon (Unknown); Patras University Hospital, Patras (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 9642
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Virus-HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIV-infected patients (Other): HIV-infected patients >= 45 years with 2 or more CV risk factors currently on ART and HIV-RNA < 50 copies >= 12 months (one blip allowed) As part of this research, three additional tubes of blood (EDTA) will be taken from patients (21 mL) during blood tests performed as part of a scheduled consultation for the management of their pathology
  Interventions: Biological: blood test

INTERVENTIONS:
Biological: blood test — Additional 21 ml of blood will be collected

SUMMARY:
HIV-infected patients with intermediate-high risk have a high prevalence of CAD and a substantial proportion of obstructive CAD. Degree of stenosis is associated with immunoactivation (lymphocyte and monocyte) and microbial translocation

DETAILED DESCRIPTION:
A hallmark of HIV infection is a state of global immune activation that is only partially restored under highly active antiretroviral therapy. Apart from immune deficiency and impaired immune restoration, this chronic immune activation may result via various mechanisms in non-AIDS linked morbidities such as atherosclerosis. Coronary artery disease (CAD), especially myocardial infarction (MI), is the leading cause of death in Europe [Eurostat 2013]. Cardiovascular deaths are responsible for 8% of deaths among HIV-infected patients in France and for 15% of deaths among HIV-infected patients in US [Lewden C JAIDS 08, Palella FJ JAIDS 06]. Multiple cohort studies have shown that HIV-infected patients are at a higher risk of myocardial infarction than the general population [Triant VA J Clin Endocrinol 07, Freiberg MS JAMA Intern Med 13] and there is some evidence that HIV-infected patients have a 38% greater risk of mortality from MI than controls [Pearce D AM J Cardiol 12].

Several tools for cardiovascular risk stratification are available but current risk scores seem to underestimate this risk in HIV-infected patients. Indeed, a significant proportion of cardiovascular events occur in subjects with none or few risk factors. A European study comparing first episode of MI among HIV-infected patients with uninfected controls showed that 40% had none or only one traditional cardiovascular risk factor [Boccara F Eur Heart J 11]. Another study in general population demonstrates that almost 50% of patients with a MI had no previous history of coronary symptoms [Tunstall-Pedoe H Circulation 96].

The true prevalence of CAD in asymptomatic HIV-infected patients is unknown. Older studies performed in tissue samples from deceased patients demonstrated 3-times greater odds of having obstructive CAD in HIV-infected patients compared with non-infected controls after controlling for age and sex [Micheletti RG Cardiovasc Pathol 09]. A recent meta-analysis shows that the prevalence of coronary stenosis and calcified coronary plaques is similar in comparison with non-HIV age and sex-matched controls but HIV-infected patients have a 3-fold higher prevalence of non-calcified coronary plaques [D'Ascenzo Atherosclerosis 15].

CAD severity detected by coronary computed tomographic angiography (CCTA) is associated with cardiac death or MI and all-cause mortality [Habib F Int J Cardiol 12]. 64 slice or greater CCTA is reported to have a sensitivity of 93 to 97% and specificity of 80 to 90% compared to standard coronary angiography [Fihn SD J Am Coll Cardiol 12]. There is a high correlation between CCTA and invasive coronary angiography in the determination of CAD extent and severity [Miller JM N Engl J Med 08].

Whether routine CCTA screening in high-risk populations can effect changes in treatment (such as pre-emptive coronary revascularization or more aggressive medical therapy) remains unproven. The 2013 AHA guidelines about stable ischemic heart disease states that either stress test or anatomic imaging in higher-risk individuals may be appropriate [J Am Coll Cardiol 14].

Few studies using CCTA have been performed in HIV-infected patients and none of these have been done in intermediate-high risk populations. Most of theses studies have shown an increased prevalence of non-calcified plaques in HIV-infected men (59% vs. 34%) compared with controls non infected with similar CVRF [Lo J AIDS 10, Post W Ann Intern Med 14]. There is some inconsistent data regarding clinical variables associated with coronary stenosis. Meanwhile CD4 nadir, use or ART for more than 10 years and detectable viral load were independently associated with coronary stenosis > 50% in the MACS cohort study [Post W Ann Intern Med 14], another study among African-Americans with HIV only cardiovascular risk factors and cocaine use were associated with coronary stenosis [Lai S Clin Infec Dis 08] Although the epidemiology and pathogenesis of HIV associated cardiovascular disease are complex and controversial we know that the risk of cardiovascular events is higher in untreated than treated HIV infection, probably because inflammation is increased in untreated infection. Recent data have raised interest in the role of Monocytes/macrophages in HIV-associated cardiovascular disease. Increased levels of monocytes activation markers such as sCD14 and sCD163 are associated with increased all-cause mortality and HIV progression, as well as more rapid progression of carotid atherosclerosis, aortic inflammation and non-calcified coronary plaque [Kelesidis JID 12, Subramanian S, JAMA 12, Burdo JID 11]. There is some evidence that monocyte profile in untreated HIV infection mirrors those with acute coronary syndrome [Funderberg N Blood 12] and circulating monocytes CD16+ were associated with coronary artery calcium progression in the SUN cohort [Baker AIDS 14]. Data from the MACS cohort showed that elevated levels of monocyte activation markers (sCD163, sCD14 and CCL2) in HIV-infected men were associated with CAC and coronary artery stenosis [Mc Kibben RA J Infec Dis 15]. None of these studies have been performed in cardiovascular high-risk virologically suppressed patients.

HIV infection causes dramatic damage to the gastrointestinal (GI) tract that includes substantial disruption of gut microbiota composition with presence of microbes at higher pathogenic potential compared to less agressive indigenous organisms, and massive loss of gut-residing CD4+ T-cells (Brenchley NAT MED 2006, Gori J Clin Microbiol 2007, Douek Annu Rev Med 2009). Thus, a substantial breach of the anatomo-functional GI barrier occurs, with progressive failure of mucosal immunity and leakage into the systemic circulation of bacterial by-products, such as lipopolysaccharide (LPS) and bacterial DNA fragments which contribute to immune activation even in patients with good virologic control (Brenchley Nature Med 2006, Jiang JID 2009, Ferri JID 2010, Estes PLoS Pathog 2010). Microbial translocation is defined as the transfer of gut derived microbes and/or microbial products to systemic circulation without overt bacteremia. Different markers may be used in order to evaluate this phenomenon: 16S DNA, LPS or its soluble receptor LBP (LPS Binding Protein), sCD14 and I-FAB. These markers are not redundant because they describe different aspects of microbial translocation. For instance 16S DNA measures global presence of microbes in plasma, while LPS increase is mainly driven by gram negative bacteria.

Persistent immune activation has been implicated in risk of cardiovascular disease in HIV infection and should receive as much attention as traditional CVD risk factors and ART (Currier AIDS 2005, Friis-Moller NEJM 2003, Subramanian JAMA 2012, Shaked Arterioscler Thromb Vasc Biol 2014, Kelesidis JID 2012). There are some reports associating LPS with subsequent cardiovascular disease in HIV-infected patients (Pedersen 2013 Kelesidis JID 2012). Increased levels of CD14s that persist in some treated HIV have been associated to an increased all-cause mortality and HIV progression, as well as more rapid progression of carotid atherosclerosis (Kelesidis T at al CROI 2012 Seattle). sCD163, a marker of monocyte and macrophage activation, has been significantly correlated with aortic inflammation (Subramanian S, JAMA 2012). Associations of one or more markers of microbial translocation with characteristics of coronary injuries (stenosis, volume, mass and type of coronary plaques) have not yet been studied.

ELIGIBILITY:
Inclusion Criteria:

HIV-infected patients >= 45 years with 2 or more CV risk factors currently on ART HIV-RNA < 50 copies >= 12 months (one blip allowed) Asymptomatic regarding cardiac symptoms (chest pain, syncope, dyspnea) Stable ART for more than 6 months

Exclusion Criteria:

Previous CV event (MI, stroke, unstable angina, CABG) Atrial fibrillation Chronic kidney disease [eGFR < 60ml/min MDRD or CKD-Epi) Unstable liver disease History of IV contrast allergy Chronic inflammatory disorders apart from HIV

Ages: 48 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-01-05 (Actual); Study Completion 2018-01-05 (Actual)

PRIMARY OUTCOMES:
coronary computed tomographic angiography (CCTA) | 1 month
  Assessment of the prevalence of obstructive coronary artery disease in patients infected with HIV and asymptomatic with a 64-slice CT coronary angiography.

SECONDARY OUTCOMES:
Lymphocyte immune activation | 1 day
  Lymphocyte immune activation (CD4+HLA-DR+, CD8+CD38+HLA-DR+)
Lymphocyte immunosenescence | 1 day
  Lymphocyte immunosenescence (CD4+CD57+, CD8+CD57+ )
Monocyte subpopulation | 1 day
  Monocyte subpopulation (CD16+ surface density) and activation markers (sCD163, sCD14, CCL2)
Microbial translocation | 1 day
  Microbial translocation (16S DNA, LBP, I-FAB and sCD14)
Inflammation | 1 day
  Inflammation (CRP, sTNFR1, IL-6, D-dimers)

CONTACTS AND LOCATIONS:
Overall Officials: Christina PSOMAS, Study Director — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC